CLINICAL TRIAL: NCT05287165
Title: Clinical Trial to Evaluate the Safety and Efficacy of IM96 CAR-T Cells Therapy in Patients With Advanced Digestive System Neoplasms
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YMCART9601
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Advanced Solid Tumors; Digestive System Neoplasms; Pancreatic Cancer Resectable; Colorectal (Colon or Rectal) Cancer
Keywords: Digestive System Neoplasms; Pancreatic Cancer Resectable; Colorectal (Colon or Rectal) Cancer
MeSH Terms: conditions — Digestive System Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM96 CAR-T cells (Experimental)
  Interventions: Drug: IM96 CAR-T cells

INTERVENTIONS:
Drug: IM96 CAR-T cells — treatment with anti-GUCY2C chimeric antigen receptor T-cell infusion

SUMMARY:
This is a open-label, single center to determine the efficacy and safety of IM96 CAR-T cells in Patients With Advanced Digestive System Neoplasms

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years, either sex;
* Patients with pathologically diagnosed advanced gastrointestinal cancer:Patients with metastatic colorectal cancer who have failed or cannot tolerate second-line or above standard treatment;Patients with unresectable locally advanced or metastatic pancreatic cancer who have failed or cannot tolerate first-line or above standard treatment; Patients with unresectable locally advanced or metastatic other gastrointestinal cancer (gastric cancer, esophageal cancer, small intestinal cancer, etc.) who have failed or cannot tolerate standard treatment, or have no standard treatment regimen;
* At least one measurable lesion meeting RECIST 1.1 criteria;
* Tumor tissue samples were positive for GUCY2C IHC staining;
* Estimated life expectancy >3 months;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Women of childbearing age who had a negative blood pregnancy test before the start of the trial and agreed to take effective contraceptive measures during the trial period until the last follow-up; male subjects with fertility partners agreed to take effective contraceptive measures during the trial period until the last follow-up;
* Adequate organ function;
* Volunteer to participate in this trial and sign on the informed consent.

Exclusion Criteria:

* Patients have brain metastasis；
* Patients with a history of organ transplantation or awaiting organ transplantation;
* The side effects caused by the previous treatment of the subjects did not return to CTCAE ≤1; other tolerable events determined by investigator;
* There is a large amount of serous effusion that cannot be controlled by treatment (such as pleural effusion, peritoneal effusion and pericardial effusion);
* History of autoimmune disease (eg Crohn's disease, rheumatoid arthritis, systemic lupus) within the last 2 years;
* Presence of acute or chronic graft-versus-host disease (GVHD);
* Use prohibited drugs or treatments within a specified period of time before cell collection；
* History or presence of CNS disorder, such as epilepsy, epileptic seizures, cerebrovascular disease (ischemia / hemorrhage / cerebral infarction), brain edema, reversible posterior white matter encephalopathy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, cerebral organic syndrome or mental disease;
* Chronic or active infections requiring systemic treatment, and a history of symptomatic viral infection that has not been completely cured；
* Live vaccine received within 6 weeks before the start of screening;
* Cardiac dysfunction includes: long QTc syndrome or QTc interval > 480 MS; Complete left bundle branch block, grade II / III atrioventricular block; Serious and uncontrolled arrhythmias requiring drug treatment; A history of chronic congestive heart failure with NYHA ≥ 3, and the cardiac ejection fraction was less than 50% within 6 months before screening; Cardiac valvular disease with CTC AE ≥ 3; Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, history of severe pericardial disease or other clinically significant heart diseases within 6 months before screening;
* Patients requiring anticoagulant therapy;
* Patients requiring continuous anti-platelet therapy;
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment;
* A history of malignancy other than non melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast), unless it has been disease-free for at least 3 years;
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection (UTI) and bacterial pharyngitis are permitted if the investigator evaluates that it can be controlled by treatment, they can be included in the group;
* Patients with gastrointestinal obstruction;
* Patients at high risk of hemorrhage or perforation;
* Patients were enrolled in another clinical study at the same time, unless it was an observational (non intervention) clinical study;
* In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 28 days after CAR-T cell infusion
  Incidence of treatment related AE.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 weeks after CAR-T cell infusion
  ORR, defined as the proportion of participants with a complete response or partial response, as determined by the investigator according to RECIST v1.1
Progression-free survival (PFS) | Up to 24 weeks after CAR-T cell infusion
  PFS, defined as the time from CAR-T cell infusion to the first occurrence of disease progression or death from any cause (whichever occurs first) , as determined by the investigator according to RECIST v1.1
Duration of Response (DOR) | Up to 24 weeks after CAR-T cell infusion
  DOR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to RECIST v1.1
Overall survival (OS) | Up to 24 weeks after CAR-T cell infusion
  OS , defined as the time from CAR-T cell infusion to death from any cause
Persistence of CAR-T cells (cell counts and cell percentage in peripheral blood) | Up to 24 weeks after CAR-T cell infusion
  The persistence over time of CAR T cells in the peripheral blood as determined by flow cytometry and qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China